CLINICAL TRIAL: NCT06415487
Title: A Phase 1 Multicenter Study Evaluating the Safety and Efficacy of ACE2016, an Allogeneic Anti-EGFR Conjugated Gamma Delta T Cell (gdT) Therapy in Adult Subjects With Locally Advanced or Metastatic Solid Tumors Expressing Epidermal Growth Factor Receptor (EGFR)
Brief Title: ACE2016 in Adult Subjects With Locally Advanced or Metastatic Solid Tumors Expressing Epidermal Growth Factor Receptor (EGFR)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acepodia Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE2016-001
Record Dates: First submitted 2024-04-30; First posted 2024-05-16 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cyclophosphamide; fludarabine; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ACE2016 ONLY: 1 DOSE (Experimental): ACE2016 dose escalation, monotherapy. Lymphodepleting regimen followed by escalating doses of ACE2016.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: ACE2016
- ACE2016 ONLY: 3 DOSES (Experimental): ACE2016 recommended dose, monotherapy. Lymphodepleting regimen followed by recommended dose of ACE2016.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: ACE2016
- ACE2016 AND PEMBROLIZUMAB: 3 DOSES (Experimental): ACE2016 recommended dose, in combination with pembrolizumab. Lymphodepleting regimen followed by recommended dose of ACE2016, giving in combination with pembrolizumab.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: ACE2016; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cyclophosphamide — Lymphodepleting agent
Drug: Fludarabine — Lymphodepleting agent
Drug: ACE2016 — Allogeneic gamma delta T (gdT) cell therapy
Drug: Pembrolizumab — Immune checkpoint anti-PD-1 antibody
  Arms: ACE2016 AND PEMBROLIZUMAB: 3 DOSES

SUMMARY:
ACE2016 is an off-the-shelf, allogeneic gamma delta T (gdT) cell therapy derived from healthy donors, that is under investigation for the treatment of Locally Advanced or Metastatic Solid Tumors Expressing Epidermal Growth Factor Receptor (EGFR).

The ACE2016-001 study is an open-label, Phase I, first-in-human (FIH) study that aims to evaluate the safety and tolerability, persistency, pharmacodynamics and efficacy of ACE2016 in patients with Locally Advanced or Metastatic Solid Tumors Expressing Epidermal Growth Factor Receptor (EGFR).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced unresectable or metastatic solid tumors that have failed at least two lines of therapy (one of which must be targeted therapy)
* At least one measurable lesion as defined by RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Adequate hematologic and renal, hepatic and cardiac function
* Oxygen saturation via pulse oximeter ≥92% at rest on room air

Exclusion Criteria:

* Prior treatment with a genetically modified cell therapy product targeting EGFR
* History of allogeneic transplantation
* Subjects with active CNS metastases
* History or presence of clinically relevant Central Nervous System (CNS) disorder (e.g. epilepsy)
* Clinically significant active infection
* Human Immunodeficiency Virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* History of malignancies with the exception of certain treated malignancies with no evidence of disease.
* Primary immunodeficiency disorder
* Pregnant or lactating female
* Any medical, psychological, familial, or sociological conditions that, in the opinion of the Investigator or Sponsor Medical Monitor, would impair the ability of the subject to receive study treatment or comply with study requirements, including understanding and rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs, AESIs, Grade 3 or higher TEAEs, TEAEs considered related to ACE2016, TEAEs resulting in death, SAEs, related SAEs, and TEAEs leading to treatment discontinuation will be summarized by cohort | 1 year
Change from baseline in clinical laboratory tests results | 1 year
  Number of subject with change from baseline clinical significant lab findings by cohort (descriptive)
Change from baseline in vital signs results | 1 year
  Number of subjects with change from baseline clinical significant vital signs findings by cohort (descriptive)
Recommended Dose (RD) | 1 year

SECONDARY OUTCOMES:
Persistence of ACE2016 before and after administration | 1 year
  Half-life of ACE2016
Measure of anti-ACE2016 antibodies after administration | 1 year
  Titration of anti-ACE2016 antibodies after administration
Objective Response Rate (ORR) | 1 year
  Proportion of subjects assessed as having a complete response (CR) or partial response (PR) according to RECIST v1.1
Disease Control Rate (DCR) | 1 year
  Number of subjects with a complete response (CR), partial response (PR) or stable disease (SD) as defined by RECIST v1.1
Duration Of Response (DOR) | 1 year
  Duration (time) from the first tumor assessment showing response per RECIST v1.1 to the time of disease progression or death.
Progression Free Survival (PFS) | 1 year
  Duration (time) from first ACE2016 cell infusion to first documentation of disease progression per RECIST v1.1 or death

OTHER OUTCOMES:
Pharmacodynamics of ACE2016 | 1 year
  Change from baseline IL2,6,8,10 IFN TNF, and change in TBNK cell subsets.
gdT infiltration in tumor mass | 1 year
  Optional biopsy to examine gdT cell infiltration

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - University of California San Diego, San Diego, California
  - SCRI Denver Drug Development Unit, Denver, Colorado
  - Sarah Cannon Research Institute (SCRI) Oncology Partners, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
- Taiwan (5):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Chang Gung Medical Foundation Linkou, Taoyuan, Guishan District
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City, Zhonghe District
  - Mackay Memorial Hospital Taipei, Taipei, Zhongshan District
  - Taichung Veteran General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No